CLINICAL TRIAL: NCT06771349
Title: Assessment of Recurrence Rate After Sigmoidopexy for Acute Sigmoid Volvulus
Brief Title: Treatment of Sigmoid Volvulus
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xiaomei Jiang, Resident Physician, Sichuan University
Other Study IDs: 2023-1601
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Sigmoid Volvulus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- sigmoidopexy group: patients who underwent sigmoidopexy
  Interventions: Procedure: sigmoidopexy
- sigmoidectomy group: patients who underwent sigmoidopexy without resection

INTERVENTIONS:
Procedure: sigmoidopexy — Both Sigmoidectomy and sigmoidopexy can be used for the treatment of sigmoid volvulus. The former is the treatment of sigmoid volvulus by removing a portion of the sigmoid colon, and depending on the patient's condition, a bowel reconstruction or anastomosis may be performed to reattach the healthy bowel segment. The procedure may result in long-term bowel changes and may even require an stomy. sigmoidopexy is a procedure that immobilizes the sigmoid colon to the abdominal wall or pelvic structure, preventing it from twisting again.
  The goal of sigmoidectomy is primarily to remove damaged or necrotic portions of the sigmoid colon and to treat complications resulting from sigmoid volvulus, especially when the volvulus results in intestinal necrosis, ischemia, or other serious complications. The goal of sigmoidopexy is to prevent the sigmoid from re-twisting by immobilizing the sigmoid, and it is suitable for those cases of sigmoid torsion without severe ischemia or necrosis.
  Groups: sigmoidopexy group

SUMMARY:
Colonic volvulus, where part of the colon twists, is a significant cause of large bowel obstruction, representing 15% of cases, second only to cancer and diverticulitis. Acute sigmoid volvulus (SV), which affects the sigmoid colon, is the most common type, with morbidity rates ranging from 6% to 42% and mortality varying from 7% to 90%. The incidence of SV varies globally, being more common in regions such as Africa, Ethiopia, Australia, and East Asia, where it can account for up to 50% of bowel obstructions.

SV often presents as partial or complete obstruction and can lead to severe complications such as ischemia, necrosis, and perforation, especially in older patients. The primary treatment goals are relieving the obstruction, reducing pressure, and correcting the twist. According to the World Society of Emergency Surgery (WSES), endoscopic decompression is recommended for patients without infection, perforation, or hemodynamic instability. However, surgery is necessary if decompression fails, with options including sigmoidopexy, sigmoidectomy, or colostomy. Sigmoidopexy is less invasive but has a higher recurrence rate, while sigmoidectomy, though riskier, may reduce recurrence and improve long-term survival.

This retrospective study aims to compare the outcomes of sigmoidopexy and sigmoidectomy in patients with acute SV undergoing emergency surgery at West China Hospital, Sichuan University, over a 14-year period. The primary outcome is the recurrence rate of SV, with secondary outcomes including 30-day mortality and morbidity (complications).

DETAILED DESCRIPTION:
Introduction:

Colonic volvulus, a significant cause of large bowel obstruction, occurs when a segment of the colon twists, obstructing normal bowel function. Among the different types of colonic volvulus, acute sigmoid volvulus (SV) is the most common, with a high incidence in certain regions, such as the "twist belt" in Africa, Ethiopia, East Asia, and Australia, where its frequency can exceed 50%. SV frequently presents as either partial or complete bowel obstruction, leading to ischemia, necrosis, and potential perforation if untreated. The morbidity and mortality associated with SV are substantial, particularly in elderly patients. Prompt management is crucial to reduce complications and improve patient outcomes.

Treatment Approaches:

The primary goal of treatment is to relieve the obstruction and address the twisted portion of the colon. The World Society of Emergency Surgery (WSES) recommends endoscopic decompression for patients without signs of severe infection, perforation, or hemodynamic instability. If decompression fails, or if necrosis is present, surgical intervention is necessary. Surgical options include sigmoidopexy, sigmoidectomy, mesenteroplasty, or colostomy. Sigmoidopexy is less invasive but carries a higher risk of recurrence, whereas sigmoidectomy, though more complex, may reduce recurrence and improve long-term survival.

Despite various treatment options, the optimal approach remains unclear due to inconsistencies in the existing literature. This study compares two commonly used surgical methods-sigmoidopexy and sigmoidectomy-to assess their outcomes in terms of SV recurrence, complications, and overall survival.

Methods:

This retrospective study reviewed patients who underwent emergency surgery for acute SV at West China Hospital, Sichuan University, between April 2009 and August 2023. The hospital, a major medical center in Chengdu, China, treats thousands of emergency cases annually. Ethical approval was obtained from the hospital's Ethics Review Board, and informed consent was waived due to the study's retrospective nature.

Inclusion Criteria:

Adults with acute symptoms of intestinal obstruction. Acute SV diagnosis confirmed by CT or surgery. First emergency surgery for acute SV at the hospital.

Exclusion Criteria:

Torsion of parts of the colon other than the sigmoid. Non-surgical management of acute SV or treatment at another institution. Conditions such as bowel perforation or unrelated obstructions. Patients unable to undergo surgery due to poor health.

Primary Outcome:

Recurrence rate of SV after sigmoidopexy or sigmoidectomy.

Secondary Outcomes:

30-day mortality and morbidity, assessed by the Clavien-Dindo classification of complications.

Data Collection:

Data were extracted from the hospital's medical records and supplemented by telephone follow-up with patients or their families. Information collected included:

Demographic details (age, gender, symptoms). Medical history (comorbidities, previous surgeries). ASA score, BMI, surgery details, and post-operative recovery. Surgical duration, hospital stay length, complications, and follow-up data.

Statistical Analysis:

Statistical analysis was conducted using R software (version 4.3.3). Continuous variables were assessed for normal distribution and expressed as means ± standard deviation or medians with ranges. Categorical variables were presented as percentages. For comparing continuous variables, Student's t-test or Mann-Whitney U test was used. For categorical data, Chi-square or Fisher's exact test was applied. A P-value of < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients presenting with symptoms of acute intestinal obstruction.
2. Diagnosis of acute SV confirmed by the typical "whirl sign" on computed tomography (CT) or laparotomy.
3. First emergency surgery for acute SV performed at our institution.

Exclusion Criteria:

1. Torsion of intestinal segments other than the sigmoid.
2. Patients diagnosed with "acute SV" but treated conservatively or operated on at another hospital.
3. Concurrent conditions such as non-SV-related bowel perforation or obstruction.
4. Patients with severe overall states not amenable to surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients (≥18 years) who underwent emergency surgery for acute sigmoid volvulus (SV) at West China Hospital, Sichuan University, between April 2009 and August 2023. Inclusion criteria: (1) Adults presenting with acute intestinal obstruction symptoms, (2) Confirmed diagnosis of acute SV via CT imaging (whirl sign) or intraoperative findings, (3) First emergency surgery for acute SV, either sigmoidopexy or sigmoidectomy. Exclusion criteria: (1) Torsion of bowel segments other than the sigmoid colon, (2) Prior conservative or surgical treatment for acute SV at another institution, (3) Concurrent bowel conditions unrelated to SV (e.g., perforation), (4) Severe comorbidities unfit for surgery. Patients who met all inclusion criteria and none of the exclusion criteria were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
To determine the recurrence rate of SV following sigmoidopexy or sigmoidectomy. | between April 2009 and August 2023
  The recurrence rate is the number of cases in which a patient has a recurrent torsion of the sigmoid colon after surgical treatment, as a proportion of all patients who undergo surgical treatment, and is usually calculated by the following equation: Recurrence rate = the number of patients with recurrence of sigmoid volvulus after surgery /the total number of patients who underwent surgery ×100%

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Gastrointestinal Surgery, Department of General Surgery, West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared publicly. However, upon request, the corresponding author can provide access to the data for specific research purposes, subject to approval.